CLINICAL TRIAL: NCT05486585
Title: Internet-delivered Psychological Treatment of Functional Gastrointestinal Disorders in Youth: the Impact of Negative Illness Understanding and Parental Illness Worries
Brief Title: i-CBT Functional Gastrointestinal Disorders in Youth: the Impact of Negative Illness Understanding and Parental Illness Worries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Skovslund Nielsen, PhD-Student, Medical doctor, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGID pilot test
Record Dates: First submitted 2022-07-06; First posted 2022-08-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-01

CONDITIONS: Functional Abdominal Pain Syndrome; Functional Gastrointestinal Disorders; Irritable Bowel Syndrome
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: An open end pilot study including 30 children and 30 adolescents and their parents (n=60)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children and Adolescents (Experimental): 30 children aged 8-12 years old and their parents, 30 adolescents aged 13-17 years old and their parents
  Interventions: Other: Internet delivered cognitive behavioural therapy for functional gastrointestinal disorders

INTERVENTIONS:
Other: Internet delivered cognitive behavioural therapy for functional gastrointestinal disorders — The offered treatment will be the Danish versions of the Swedish i-CBT programs for children. The child i-CBT program consists of 10 modules for the child and 10 for parents. The adolescent i-CBT program consists of 10 modules for the adolescent and 5 modules for the parents. Child and adolescents modules compose of exposure exercises for symptoms, behavioural analyses and affect labelling and are adjusted for the specific age group. Parent modules aim at supporting parents in helping their child to engage in the challenging exposure exercises. The family needs to select one parent to participate in the parent program. The participants will be expected to use approximately 4 hours per week. The programs will be delivered over ten weeks, and therapist support will be provided on a weekly basis.

SUMMARY:
The aim of the current study, embedded in The Danish FGID Treatment Study, is to test Danish versions of Swedish i-CBT programs for children and adolescents with FGID in a Danish clinical context and to further evaluate the presence and impact of important psychological and parental factors.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGID) are common among children and adolescents. They affect quality of life, cause functional disability, school absence and high health care use.

Parental behavior can significantly influence the young person's perception of bodily symptoms, which are thought to be part of development and maintenance of symptoms FGID. So are cognitive biases which are distortions in attention, memory and interpretation.

The programs involve both the youth and their parents, which provides a unique possibility, to examine illness-related cognitive biases and the effectiveness of graded exposure in youths with FGID with an additional focus on parental distress and illness worries for treatment adherence and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Child age: 8-12 years, adolescents: 13 - 17 years
* A primary diagnosis according to the ROME-IV criteria of one of the FGID sub-types: Irritable bowel syndrome (IBS) or functional abdominal pain not-otherwise-specified (FAP-NOS)
* The diagnosis should be documented by their regular physician in the somatic setting, and recommended routine medical investigations should be evaluated as normal or without clinical significance (include growth; blood samples including TSH, total IgA, IgA tissue transglutaminase, complete blood count, C-reactive protein analysis, liver enzymes; and fecal calprotectin)
* Stable dosage of FGID-related medication such as laxatives, anti-diarrheal medication or pain-modulating psychopharmacological medication during the past month.

Exclusion Criteria:

* Another disease that explains the symptoms;
* Severe psychiatric or social problems (e.g., high level of suicidal ideation or ongoing abuse);
* Ongoing psychological treatment;
* Insufficient language or computer skills (patients and parents);
* Severe family problems (e.g. child abuse, parental substance abuse or severe psychiatric illness, ongoing custody fight)
* School absence of more than 40% over the past month.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in gastrointestinal symptoms assessed by PedsQL Gastro Symptom Scales | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)]
  The self-report questionnaire revised version of PedsQL Gastro Symptom Scales, with 9 items. Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Change in gastrointestinal symptoms rated by parents assessed by PedsQL Gastro Symptom Scales | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)]
  The parent-report questionnaire revised version of PedsQL Gastro Symptom Scales, with 9 items. Answered on a 5 point scale from 0 ("never") to 4 ("almost always)

SECONDARY OUTCOMES:
Changes in cognitive biases in interpretation and memory of stimuli related to gastrointestinal themes, leisure and school: Picture Task. | At baseline and 10-weeks of treatment (end of treatment)
  Online experimental task with a picture task, with 15 pictures rated on emotional valence (0 negative, 100 positive), physical reaction (1 nota at all, 7 very much) and relatability to own life (1 not at all, 7 very much). Pictures are then recalled and rated on emotional valence (0 negative, 100 positive) and physical reaction (1 nota at all, 7 very much). Lastly pictures are recognised from unfamiliar pictures and rated on difficulty (1 not at all, 7 very much) and confidence (1 not at all, 7 very much).
Changes in cognitive biases in interpretation and memory of stimuli related to gastrointestinal themes, leisure and school: Health Norms sorting Task. | At baseline and 10-weeks of treatment (end of treatment)
  Online experimental task with FGID-specific version of the Health Norms Sorting Task, Participants sort 20 words as healthy or no longer healthy, recall as many words as possible and lastly recognise from previously unfamiliar words while rating on difficulty (1 not at all, 7 very much) and confidence (1 not at all, 7 very much).
Changes in Quality of life assessed by the Pediatric Quality of Life Inventory | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The self-report questionnaire Pediatric Quality of Life Inventory 8-12-year version for children, 13-18-year version for adolescents. 23 items, Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Changes in Quality of life rated by parents assessed by Pediatric Quality of Life Inventory | Time Frame: At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The parent-report questionnaire Pediatric Quality of Life Inventory for parents, (Parent report for children aged 8-12 years, and parent report for adolescents aged 13-17 years) . 23 items, Answered on a 5 point scale from 0 ("never") to 4 ("almost always)
Changes in Pain intensity measured by the self-report rating scale, Faces pain scale, revised | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The scale consists of 6 faces representing least to most pain, and each face is connected to a number from 0 (no pain)
  - 10 (most pain),
Changes in Pain intensity rated by parents Measured by the parent-report rating scale, Faces pain scale, revised | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)]
  The scale consists of 6 faces representing least to most pain, and each face is connected to a number from 0 (no pain)
  - 10 (most pain),
Changes in Overall symptom load measured by the self-report questionnaire Children somatization inventory , short (CSI) | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consist of 24 items Answered on a 5 point scale from 0 ("not at all") to 4 ("a whole lot")
Changes in Overall symptom load rated by parents measured by the parent-report questionnaire Children somatization inventory (parent report), short | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consists of 24 items Answered on a 5 point scale from 0 ("not at all") to 4 ("a whole lot")
Changes in Depression symptoms measured by the self-report questionnaire Mood and Feelings Questionnaire short | At baseline, 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consists of 13 items, answered on a 3 point scale: not true / sometimes true / true
Changes in General Anxiety symptoms measured by the self- report questionnaire Spence Children Anxiety Scale short | At baseline, 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A 19 item-questionnaire answered on a 4 point scale from 0(never) to 3 (always)
Changes in General Anxiety rated by parents, Measured by the parent- report questionnaire Spence Children Anxiety Scale short, parent report | At baseline, 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)]
  A 19 item-questionnaire answered on a 4 point scale from 0(never) to 3 (always)
Changes in Specific Gastrointestinal Anxiety, Measured by the self-report questionnaire Visceral Sensitivity Index -Short | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A 7 item-questionnaire answered on a 5 point scale from 0 (don't agree at all) to 5 (totally agree)
Changes in Avoidance and control behaviour measured by the self-report questionnaire irritable bowel syndrome behavioural response questionnaire | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A 11 item-questionnaire answered on a 7 point likert scale from 1(never) to 7(always)
Changes in Illness perception Measured by the self-report questionnaire Brief Illness perception Questionnaire | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A questionnaire with 11 items answered on a scale from 0 - 10
Changes in Illness perception rated by parents, measured by the parent-report questionnaire Illness perception regarding child's symptoms Questionnaire | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  A questionnaire with 11 items answered on a scale from 0 - 10
Changes in Illness worry Measured by the self-report questionnaire Childhood Illness Attitude Scale | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The fear-factor domain of the questionnaire is used, it consists of 11 items, answers: never, sometimes or always
Changes in Acceptance, measured by the self-report questionnaire Chronic pain Acceptance Questionnaire -adolescents | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Two items from the self-report questionnaire Chronic pain Acceptance Questionnaire -adolescents are used. 2 selected items, answered on a 5-point scale from 0 (never true) to 4 (always true)
Changes in PARENTAL Illness Worry measured by the self-report The Health Anxiety by Proxy Scale (HAPYS) questionnaire | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Parental illness worry for their child, measured by the self-report The questionnaire covers 26 items about health anxiety by proxy, rated on a five-point scale (from "not at all"/"never" to "a whole lot"/"most of the time"). And five items about the impact of the worries rated on a four-point scale (from "no" to "yes, severely").
Changes in PARENTAL Emotional distress measured by the self-report questionnaire Symptom Check List (SCL-8) | At baseline, after 5 weeks of treatment (mid-treatment), after 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  The questionnaire consists of 8 items answered on a 5 point scale from 0 (not at all) to 4 (a whole lot)
Changes in Adult Response to Child's Symptoms - PARENTS by the self-report questionnaire Adult Response to Children's Symptoms | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Protect and Monitor scale from the the questionnaire Adult Response to Children's Symptoms used, 15 items answered on a 5 point scale from 0(never) to 4 (always)
Changes in School absence / Work absence parent | At baseline, 5 weeks of treatment (mid-treatment), 10 weeks of treatment (end-treatment) and 3-months after treatment (follow-up)
  Question about Hours / Days missed from school/work last month. Parental report for children aged 8-12 years, self-report for adolescents aged 13-17 years, self-report for parents

OTHER OUTCOMES:
Treatment satisfaction by the self-report questionnaire Modified Experience of Service Questionnaire Modified Experience of Service Questionnaire | At 10 weeks of treatment (End of treatment)
  10 items rated either true, partly true, not true or don't know and 3 open end questions
Adverse events | At 10 weeks of treatment (End of treatment)
  Open end questions. Parents to children aged 8-12 years will answer on behalf of their children and adolescents aged 13-17 years will answer themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ulrikka Rask, Professor, MD, PhD, Study Chair — Aarhus University and Aarhus University Hospital, Child and Adolescents Psychiatry
Locations (1):
- Aarhus University and Aarhus University Hospital, Child and Adolescents Psychiatry, Aarhus, Denmark

REFERENCES:
- [Derived] Skovslund Nielsen E, Kallesoe K, Bennedsen Gehrt T, Bjerre-Nielsen E, Lalouni M, Frostholm L, Bonnert M, Rask CU. Trajectories of Change, Illness Understanding, and Parental Worries in Children and Adolescents Undergoing Internet-Delivered Cognitive-Behavioral Therapy for Functional Abdominal Pain Disorders: Protocol for a Single-Case Design and Explorative Pilot Study. JMIR Res Protoc. 2025 Jan 7;14:e58563. doi: 10.2196/58563. PMID 39773759